CLINICAL TRIAL: NCT07184814
Title: Clinical Features and Prognosis of Takayasu's Arteritis With Pulmonary Arteries Involvement
Acronym: CAPTAIN
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Wanmu Xie, Director, Department of Integrative Pulmonary Medicine, China-Japan Friendship Hospital
Other Study IDs: 2022-NHLHCRF-LX-01-01-02
Record Dates: First submitted 2025-09-10; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Takayasu Arteritis With Pulmonary Artery Involvement; Pulmonary Arterial Hypertension Associated With Connective Tissue Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAK-PAI group

SUMMARY:
The purpose of this study is to identify the clinical features, management pattern and long-term outcomes of patients with pulmonary arteries involvement in Takayasu's arteritis (TAK-PAI).

DETAILED DESCRIPTION:
The present study intends to conduct a prospective analysis of the clinical data in TAK patients in order to:

1. describe the clinical characteristics and current status of multimodal treatment in patients with TAK-PAI, thereby enhancing the understanding of TAK-PAI;
2. to investigate the risk factors for mortality in patients with TAK-PAI, so as to promote early intervention and reduce mortality.
3. explore factors associated with pulmonary hypertention (PH) in patients with TAK-PAI, so as to facilitate the early identification of patients who may develop PH.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized between Jan 1, 2016 and Dec 31, 2026
* Diagnosed with TAK according to the modified Ishikawa criteria and/or 1990 American College of Rheumatology criteria and/or 2022 ACR/EULAR criteria
* Diagnosed with pulmonary artery involvement using computed tomography pulmonary angiography or transcatheter pulmonary angiography
* Patients without aortic or primary branch involvement who nonetheless exhibited both clinical features and computed tomography-confirmed evidence of pulmonary artery involvement (PAI), after exclusion of other diseases causing pulmonary artery stenosis or occlusion

Exclusion Criteria:

* Patients with PAI caused by non-TAK diseases such as other types of vasculitis, fibrosing mediastinitis, pulmonary artery sarcoma, pulmonary sarcoidosis or chronic thromboembolic pulmonary hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: TAK patients hospitalized at the China-Japan Friendship Hospital, Beijing Anzhen Hospital and Beijing Chaoyang Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause death | At 3 months, 6 months, and annually thereafter following enrollment, until December 31, 2026.

SECONDARY OUTCOMES:
Six-minute walk distance | At 3 months, 6 months, and annually thereafter following enrollment, until December 31, 2026
WHO functional class | At 3 months, 6 months, and annually thereafter following enrollment, until December 31, 2026.
N-terminal pro-brain natriuretic peptide level | At 3 months, 6 months, and annually thereafter following enrollment, until December 31, 2026

OTHER OUTCOMES:
Mean pulmonary arterial pressure assessed by right heart catheterization | At 3 months, 6 months, and annually thereafter following enrollment, until December 31, 2026.
  Hemodynamic parameters assessed by right heart catheterization in patients with pulmonary hypertension.
Pulmonary vascular resistance assessed by right heart catheterization | At 3 months, 6 months, and annually thereafter following enrollment, until December 31, 2026.
  Hemodynamic parameters assessed by right heart catheterization in patients with pulmonary hypertension.
Cardiac output assessed by right heart catheterization | At 3 months, 6 months, and annually thereafter following enrollment, until December 31, 2026.
  Hemodynamic parameters assessed by right heart catheterization in patients with pulmonary hypertension.
Cardiac index assessed by right heart catheterization | At 3 months, 6 months, and annually thereafter following enrollment, until December 31, 2026.
  Hemodynamic parameters assessed by right heart catheterization in patients with pulmonary hypertension.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship hospital, Beijing, Beijing Municipality, China